CLINICAL TRIAL: NCT07014293
Title: Increasing Resiliency Among Early Post-Treatment Lymphoma Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Giselle K. Perez Lougee, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 25-161; RSGHE-24-1325325-01-CTPS (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma
Keywords: coping; psychosocial intervention; survivorship; resilience
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Other): Participants randomized to EUC will be referred to their site social work team. This most closely resembles the real-world care available to survivors on an outpatient basis. It is an enhanced version of usual care because proactive identification and referral of posttreatment survivors is not routinely done.
  Interventions: Other: Enhanced Usual Care
- SMART3RP-Lymphoma (Experimental): Participants will participate in 8 weekly group sessions, delivered virtually. The intervention components include: 1. Eliciting the relaxation response (RR) involves sustained mental focus with an attitude of open receptive awareness. 2. CBT to improve stress management involves increasing awareness and identification of the components of one's stress response (negative thoughts, emotions, physical reactions, behaviors, and relational) and learning skills at each session to alter these components (e.g., cognitive restructuring). 3. Positive psychology strategies to achieve growth enhancement focus on utilizing techniques and skills to promote positive growth. Skills focus on increasing social support, positive affect, and compassion.
  Interventions: Other: SMART3RP-Lymphoma

INTERVENTIONS:
Other: Enhanced Usual Care — Participants will receive a singleevaluation with a site social worker along with a list of mental health, social or community resources . This most closely resembles the real-world care available to survivors on an outpatient basis, however, we call this enhanced usual care since proactive identification and referral of posttreatment survivors is not routinely done.
  Arms: Enhanced Usual Care
Other: SMART3RP-Lymphoma — The intervention components include: 1. Eliciting the relaxation response (RR) involves sustained mental focus with an attitude of open receptive awareness. 2. CBT to improve stress management involves increasing awareness and identification of the components of one's stress response (negative thoughts, emotions, physical reactions, behaviors, and relational) and learning skills at each session to alter these components (e.g., cognitive restructuring). 3. Positive psychology strategies to achieve growth enhancement focus on utilizing techniques and skills to promote positive growth. Skills focus on increasing social support, positive affect, and compassion.
  Arms: SMART3RP-Lymphoma

SUMMARY:
The goal of this clinical trial is to learn if a mind body resilience group program can help increase lymphoma survivors' ability to cope with and manage the challenges that come with the transition into early post treatment survivorship.

DETAILED DESCRIPTION:
This is a randomized controlled trial assessing the effects of the Stress Management and Resiliency Training: Relaxation Response Resiliency-Lymphoma (SMART3RP-Lymphoma) compared to Enhanced Usual Care on 254 early post treatment lymphoma survivors. The SMART-3RP is a comprehensive, evidence-based mind body group program designed to help individuals adapt to chronic stress (i.e., increase their resilience). It understands the adjustment to chronic stress as a dynamic process, blending CBT, positive psychology and mind body tools to target key coping processes.

This trial seeks to answer the following questions:

* Will survivors randomized to SMART3RP-Lymphoma demonstrate greater improvements in coping skills when compared to survivors randomized to enhanced usual care?
* Do factors, such as age, sex, race/ethnicity, rural/urban living, socioeconomic status, impact how survivors respond to the treatment?

ELIGIBILITY:
Inclusion Criteria:

* English speaking adult (18 years or older at enrollment)
* Within 5 years of completing active, curative treatment for lymphoma (includes surgery, chemo-/immuno-/radiation therapy, or other)

Exclusion Criteria:

* Active Psychiatric or cognitive comorbidity as determined by site PI or treating clinician
* Unwilling or unable to participate using telehealth platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Coping Scores on the Measure of Current Status Scale (MOCS-A) | Baseline to 3 month follow up
  The Measure of Current Status Scale (MOCS-A) measures coping processes on 4 domains: ability to relax, recognize stress, elicit support, and restructure thoughts. It is a 13-item scale where each item is measured on a 0-4 scale.

SECONDARY OUTCOMES:
Change in Emotional Distress (anxiety and depression) based on the PROMIS-Anxiety 8a and PROMIS-Depression 8a | Enrollment to 3 month follow up
  The PROMIS-Anxiety 8a and PROMIS-Depression 8a measure anxiety symptoms and depression symptoms, respectively. The measures are 8 items, where each item is scored on a scale of 1 (Never) - 5 (Always).
Change in Physical Health (PROMIS Physical Function-8b) | Enrollment to 3 month follow up
  The PROMIS Physical Function-8b is an 8-item measure that assesses the ability to perform daily living activities. Each item is scored on a scale of 1 (Unable to do) to 5 (Without any difficulty).
Change in Quality of Life scores (Functional Assessment of Cancer Therapy (FACT-G)) | Enrollment to 3 month follow up
  The FACT-G is a 27 item measure of quality of life on 4 domains: physical, functional, emotional, and social. Each item is measured on a 0 (not at all) to 4 (very much) scale.
Change in Resilience scores (Current Experiences Scale (CES-23)) | Enrollment to 3 month follow up
  The CES-23 is a 23-item measure that assesses resilience on 6 dimensions: appreciation for life, adaptive perspectives, personal strength, spiritual connectedness, relating to others, and health behaviors. Each item is scored on a 0 (not at all) to 5 (to a very great degree) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No